CLINICAL TRIAL: NCT01273961
Title: Radiofrequency Magnetic Induction Device for Use in Non-Invasive Body Contouring
Brief Title: Study of Radiofrequency Device for Use in Non-Invasive Cosmetic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Mountain Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0310-0003
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Laxity of Skin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AuraLevée treatment — A single treatment, on day 0, on each of no more than two treatment sites, using the AuraLevée device. Treatment sites are the face, abdomen, upper arm, thigh or neck.

SUMMARY:
The purpose of this pilot research study is to collect information on the safety and effectiveness of an experimental device used to treat and improve the appearance of the skin by reducing the visibility of wrinkles and by reducing the looseness of skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 to 70 years old,
* For females, at least 9 months post-partum,
* Clinically appreciable skin laxity on the abdomen, thigh, upper arms or neck as determined by the study investigator,
* For females, post-menopausal, surgically sterilized, or using a medically accepted form of birth control for at least 3 months prior to the study,
* Apparently healthy,
* Informed consent signed by the subject.

Exclusion Criteria:

* History of skin hypersensitivity,
* Current skin disorder (e.g. keloid scarring) or infection (e.g., herpes simplex),
* Use of non-steroidal anti-inflammatory drugs within past 2 weeks,
* Suffering from hormonal imbalance which may affect weight or cellulite,
* Subjects with pacemakers, internal defibrillators or electronically, magnetically, and mechanically activated implants,
* Subjects with implanted medical prostheses (such as clips, pins or plates) proximal to the treatment site,
* The current or recent use (within the past 12 months) of isotretinoin,
* Pregnancy or breast feeding,
* Infectious diseases (such as HIV) present,
* Are a tobacco smoker,
* Insulin dependent diabetic subjects,
* Oxygen dependent subjects,
* Subjects with severe chronic illness, scleroderma, or lupus,
* Subjects with open sores or scars in the treatment region, or
* Subjects with ischemia in the treatment region.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Improvement in cosmesis | 1 and 3 months
  Improvement in cosmesis will be assessed by scoring photographs taken before and 1 and 3 months after treatment. Circumference changes will be measured and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wolfe, MD, Principal Investigator — Center for Cosmetic Surgery; Stephen Flock, PhD, Study Director — Rocky Mountain Biosystems, Inc.
Locations (1):
- Center for Cosmetic Surgery, Golden, Colorado, United States